CLINICAL TRIAL: NCT07196488
Title: Development and Exploring the Efficacy of a Dyadic Co-learning Intervention for Patients With Prostate Cancer and Their Spouses
Brief Title: Dyadic Co-learning Intervention for Patients With Prostate Cancer and Their Spouses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hui Chien, RN, PhD, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202202198B0C1002
Record Dates: First submitted 2025-09-06; First posted 2025-09-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: Prostate cancer; emotional well-being; physical symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive routine care.
- Dyadic Co-learning Intervention Group (Experimental): Participants in the experimental group will receive routine care plus an 8-week Dyadic Co-learning Intervention.
  Interventions: Other: Dyadic Co-learning Intervention

INTERVENTIONS:
Other: Dyadic Co-learning Intervention — Participants in the experimental group will receive routine care plus an 8-week Dyadic Co-learning Intervention, which will consist of three components: (1) a co-learning handbook, (2) a co-learning mobile app, and (3) professional support.
  Arms: Dyadic Co-learning Intervention Group

SUMMARY:
This study aims to help patients with prostate cancer and their spouses cope better with the challenges of cancer by learning and supporting each other together. The investigators will test an 8-week "Dyadic Co-learning Intervention," which includes weekly learning topics, a mobile app, and professional support. The goal is to improve their physical symptoms, emotional well-being, and resilience.

Participants will be randomly assigned to one of two groups. One group will receive regular care, while the other group will receive regular care plus the new co-learning program. The investigators will ask both patients and their spouses to complete questionnaires at the beginning of the study, and again at 10 and 16 weeks, to understand how the program affects their health and well-being.

DETAILED DESCRIPTION:
Objective:

To evaluate the effectiveness of a Dyadic Co-learning Intervention for patients with prostate cancer and their spouses, focusing on physical symptoms, emotional well-being, and resilience.

Study Design:

An experimental, two-group, randomized controlled design will be adopted. Participants will be recruited through convenience sampling from the urology outpatient department and inpatient wards of a hospital. Patients diagnosed with prostate cancer and their cohabiting spouses who agree to participate will provide written informed consent prior to data collection.

Procedures:

Baseline data (Time 0) will be collected using structured questionnaires. After completing the pretest assessment, patient-spouse dyads will be randomly assigned to either the intervention group or the control group in a 1:1 ratio.

The intervention group will receive routine care plus an 8-week Dyadic Co-learning Intervention, while the control group will receive routine care only.

Follow-up assessments will be conducted at the 10th week (Time 1) and the 16th week (Time 2) after the baseline to evaluate intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

1. Diagnosed with prostate cancer by a board-certified urologist.
2. Has either decided on a treatment plan or completed treatment within the past two years.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

For Spouses:

1. Must be a cohabiting spouse of the prostate cancer patient and aged 20 years or older.
2. Must have a Barthel Index score of 91 or above, indicating good functional independence.

Exclusion Criteria:

Either the patient or the spouse will be excluded if:

1. Diagnosed with another type of cancer.
2. Diagnosed with cognitive impairment or a psychiatric disorder, such as dementia, depression, or anxiety.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Family Resilience (patients and spouses) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  This study will adopt the Chinese version of the Walsh Family Resilience Questionnaire to assess family resilience in patients with prostate cancer and their spouses. The scale uses a 5-point Likert rating, ranging from 1 (Never) to 5 (Always). Total scores range from 26 to 130, with higher scores indicating greater levels of family resilience.

SECONDARY OUTCOMES:
Physical Symptoms and Distress (patients only) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  This study will use the Chinese version of the Expanded Prostate Cancer Index Composite (EPIC-26) to assess symptoms and related distress in patients with prostate cancer. The scale consists of 26 items covering four domains: urinary incontinence, urinary irritation/obstruction, bowel symptoms and distress, sexual function and distress, and vitality/hormonal function and distress. Total scores range from 0 to 100, which higher scores indicate fewer symptoms and less distress.
Fatigue (patients only) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  The Taiwanese version of the Brief Fatigue Inventory (BFI) will be used to assess the severity of cancer-related fatigue over the past 24 hours and its impact on daily life in patients with prostate cancer. The instrument consists of 9 items; each rated on an 11-point scale ranging from 0 to 10. Higher scores indicate greater fatigue severity or greater interference with daily activities.
Resilience (patients and spouses) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  he 10-item version of the Connor-Davidson Resilience Scale (CD-RISC-10) will be used to measure individual resilience among both prostate cancer patients and their spouses. Each item is scored on a scale from 0 to 4, with total scores ranging from 0 to 40. Higher scores indicate greater resilience.
Loneliness (patients and spouses) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  The Chinese version of the Loneliness Scale will be used to assess the level of loneliness in both prostate cancer patients and their spouses. The scale consists of 9 items, covering two subscales: social loneliness and emotional loneliness. Each item is scored dichotomously (0 or 1), with total scores ranging from 0 to 9. Higher scores indicate a greater sense of loneliness.
Subjective Well-Being (patients and spouses) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  The Chinese Subjective Well-Being Scale, developed specifically for Chinese populations, will be used to measure subjective well-being among patients and their spouses. The scale includes 10 items rated on a 4-point scale (0-3), with total scores ranging from 0 to 30. Higher scores indicate greater perceived well-being.
Intervention Satisfaction (patients and spouses in intervention group) | 10th weeks after the pre-test
  This questionnaire consists of five items designed to assess participants' satisfaction with the intervention program, including the mobile application, multimedia videos, handbook, and professional support. Each item will be scored on a scale from 0 to 100, with higher scores indicating greater satisfaction.

OTHER OUTCOMES:
Age (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the ages of patients and their spouses; a higher value indicates older age.
Education level (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the education levels of patients and their spouses, categorized as: elementary school, junior high school, senior high school, college/university, and graduate degree.
Religious belief (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the religious belief of patients and their spouses, categorized as: None, Buddhism, Taoism, Christianity, Catholicism, folk religion, and others.
Employment status (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the employment status of patients and their spouses, categorized as: full-time employed, part-time employed, on medical leave (retaining employment), retired, unemployed, or other.
Number of children (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the ages of patients and their spouses; categorized as none, or number of sons and daughters (self-reported).
Relationship status (Patients and Spouses) | Before the intervention (pre-test)
  The demographic information form will be used to collect the relationship status of patients and their spouses, categorized as married, single/never married, divorced, widowed, cohabiting, or remarried.
Living arrangement (Patients) | Before the intervention (pre-test)
  The demographic information form will be used to collect the living arrangement of patients, categorized as living alone, living with spouse, living with spouse and children, living with spouse and grandchildren, living with grandchildren, or other.
Cancer stage (Patients) | Before the intervention (pre-test)
  The disease-related information form will be used to collect the cancer stage of patients.
Time since diagnosis (Patients) | Before the intervention (pre-test)
  The disease-related information form will be used to collect the time since diagnosis (in months) of patients.
Most recent PSA level (ng/mL) (Patients) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  The disease-related information form will be used to collect the most recent PSA level (ng/mL) of patients.
Initial PSA level (ng/mL) (Patients) | Before the intervention (pre-test)
  The disease-related information form will be used to collect the initial PSA level (ng/mL) of patients.
Gleason score (Patients) | Before the intervention (pre-test)
  The disease-related information form will be used to collect the gleason score of patients.
Primary treatment method (Patients) | Before the intervention (pre-test)
  Primary treatment method for prostate cancer will be collected using the disease-related information form.
History of cancer recurrence (Patients) | Before the intervention (pre-test)
  The disease-related information form will be used to collect the history of cancer recurrence among patients.
Chronic disease history (Patients and Spouses) | Before the intervention (pre-test)
  Presence of comorbidities, assessed using the disease-related information form; categorized as none, or specified conditions (diabetes mellitus, asthma, gastrointestinal ulcer, glaucoma, hypertension, bronchitis, gastroesophageal reflux disease, cataract, heart disease, stroke, arthritis/degenerative joint disease, or other).
Perceived physical health status (Patients and Spouses) | Before the intervention (pre-test), and at the 10th and 16th weeks after the pre-test
  The disease-related information form will be used to collect the perceived physical health status of patients and their spouses, with higher scores indicating better perceived physical health.
Menopausal status (Spouses) | Before the intervention (pre-test)
  Menopausal status (irregular menstruation but not complete cessation), assessed using the disease-related information form; categorized as yes/no.
History of menopause (Spouses) | Before the intervention (pre-test)
  History of menopause, assessed using the disease-related information form; categorized as yes/no. For participants who responded "yes," the age at menopause (in years) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hui Chien, Principal Investigator — National Taipei University of Nursing and Health Sciences, Taipei, Taiwan.
Locations (2):
- Taiwan (2):
  - Keelung Chang Gung Memorial Hospital, Keelung
  - LinKou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Data supporting this study's findings are available from the corresponding author upon reasonable request. The data are not publicly available due to the consideration of ethics, the researchers shall maintain the privacy of the participants, and research data should be used only for academic articles.

REFERENCES:
- [Background] Lin CC, Chang AP, Chen ML, Cleeland CS, Mendoza TR, Wang XS. Validation of the Taiwanese version of the Brief Fatigue Inventory. J Pain Symptom Manage. 2006 Jul;32(1):52-9. doi: 10.1016/j.jpainsymman.2005.12.019. PMID 16824985
- [Background] Szymanski KM, Wei JT, Dunn RL, Sanda MG. Development and validation of an abbreviated version of the expanded prostate cancer index composite instrument for measuring health-related quality of life among prostate cancer survivors. Urology. 2010 Nov;76(5):1245-50. doi: 10.1016/j.urology.2010.01.027. Epub 2010 Mar 28. PMID 20350762
- [Background] Wang A, Lu J. Validation of the Chinese version of the Walsh Family Resilience Questionnaire. Fam Process. 2023 Mar;62(1):368-386. doi: 10.1111/famp.12751. Epub 2022 Feb 23. PMID 35195282
- [Background] Meng M, He J, Guan Y, Zhao H, Yi J, Yao S, Li L. Factorial Invariance of the 10-Item Connor-Davidson Resilience Scale Across Gender Among Chinese Elders. Front Psychol. 2019 May 31;10:1237. doi: 10.3389/fpsyg.2019.01237. eCollection 2019. PMID 31214071